CLINICAL TRIAL: NCT06310564
Title: A Prospective, Randomized Clinical Trial of Low and Intermediate Risk OliGometastatic ColoREctal CancEr PatieNts Treated with Stereotactic ABlative Radiotherapy: GREEN LaIT-SABR Study
Brief Title: Low and Intermediate Risk OliGometastatic ColoREctal CancEr PatieNts Treated with Stereotactic ABlative Radiotherapy
Acronym: GREENLaIT-SABR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-18
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- stereotactic ablative radiotherapy (SABR) (Experimental): SABR to all the active sites of disease (1-3 oligometastases). 3D-CRT, IMRT and VMAT techniques are allowed, but IMRT and VMAT are strongly suggested.
  Interventions: Radiation: SABR
- no SABR (No Intervention): no SABR

INTERVENTIONS:
Radiation: SABR — A biological effective dose (BED) ≥125 Gy10 should be administered when constraints to the organs at risk (OARs) are respected [10]; if not possible, a BED schedule no lower than 100 Gy10 should be administered. In compliance with these instructions, treatment schedules, total dose and fractionation will be prescribed according to the clinical practice of each participating Center. The constraints for the organs at risk will be respected according to the available data.
  In any case, biological effective dose (BED) ≥125 Gy10 should be administered when constraints to the organs at risk (OARs) are respected; if not possible, a BED schedule no lower than 100 Gy10 should be administered.
  SABR will be administered before systemic treatment start, or before starting the second systemic treatment cycle at the latest.
  Arms: stereotactic ablative radiotherapy (SABR)

SUMMARY:
This is an experimental study without drug or device, randomized, open-label, non-profit, sponsored by the IRCCS Sacro Cuore Don Calabria Hospital in Negrar, which will take place at the Department of Advanced Oncological Radiotherapy and 18 other Italian centers.

The reason for this research study is to evaluate whether stereotactic radiotherapy treatment (SABR), in addition to the systemic chemotherapy treatment foreseen by clinical practice for low-intermediate risk oligometastatic colorectal cancer, is able to:

* delay possible local recurrence and/or distant polymetastatic progression
* improve disease-free survival
* reduce side effects in the short and long term

thus inducing an improvement in the quality of life of patients suffering from this type of pathology.

Therefore, as part of this randomized study, before starting first or second line systemic therapy for his tumor, the patient will be randomized to one of the following treatment arms:

* Experimental arm: ablative stereotactic radiotherapy on all sites of oligometastatic disease (from 1 to 3 sites, performed at most within the second cycle of systemic therapy)
* Control arm: no ablative stereotactic radiotherapy to sites of oligometastatic disease

The procedure that is intended to be tested in the experimental arm is a stereotactic radiotherapy treatment on oligometastases (up to a maximum of 3 sites), with ablative dosage (effective biological dose >100 Gy), performed before the start of systemic therapy of I or II line (at most within the second cycle of the same).

It is hoped that the addition of this type of radiotherapy will increase the potential clinical benefit of the treatment in the context of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed CRC
* Low and intermediate risk oligometastatic colorectal cancer with 1 to 3 metastases, candidate to I or II line systemic treatment (Low risk: 1 to 3 metastases and cumulative tumor volume smaller than 10 cm3; Intermediate risk: 1 to 3 metastases and cumulative tumor volume bigger than 10 cm3).
* Controlled primary tumor regardless of primary surgery or primary systemic treatment
* ECOG/WHO 0-2
* Life expectancy > 6 months
* Lesions ≤ 5 cm
* Adequate organ function for the planned treatment according to local guidelines
* For patients with liver metastases: no cirrhosis or hepatitis, and evidence of adequate hepatic function (Total bilirubin level < 1.5 x institutional ULN; ALT and AST levels < 3.0 x institutional ULN, GGT and alkaline phosphatase levels < 3.0 x institutional ULN; INR and APTT levels < 1.5 x institutional ULN, Albumin > 2.5 mg/dL)
* For patients with liver metastases: unresectable liver metastases (assessed by a surgeon, preferably hepatobiliary) or refusal of liver surgery before study screening.
* If childbearing potential, willing to use an effective form of contraception throughout the duration of the study
* Signed informed consent and willingness to follow the trial procedures

Exclusion Criteria:

* Age < 18 years
* Brain metastases
* Having more than 3 metastases
* Malignant pleural effusion or ascites
* Unable to undergo imaging by either CT scan or MRI
* Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, neurological conditions, physical examination or laboratory findings) that may interfere with the planned treatment or affect patient compliance.
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2031-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS). | 7 years
  PFS is defined as the time between randomization to the radiological evidence of disease progression.
  For patients with a PFS event, PFS will be calculated as the time interval from the date of randomization to the date of first objective evidence of disease progression or death from any cause, whichever occurs first.
  For patients without a PFS event, PFS will be censored at the date of the last radiographic assessment prior to the date of study end.

SECONDARY OUTCOMES:
Time to the polymetastatic conversion (tPMC) | 7 years
  tPMC will be defined as the time between randomization to the date of radiological occurrence of >5 new metastases. For patients without a tPMC event, time to tPMC will be censored at the date of the last radiographic assessment prior to the study end date.
Local control (LC): the time between randomization to the date of radiological development of local progression after SABR. | 7 years
  For patients without LC, time to LC will be censored at the date of the last radiographic assessment prior to the study end date.
Overall survival (OS) | 7 years
  OS will be defined as the time between randomization to the date of death or last follow-up. For patients who are alive at the time of the study end date, OS time will be censored on the last date the patient is known to be alive or the study end date, whichever occurs first.
Time to start of the next systemic treatment line (NEST) | 7 years
  For patients without a NEST, time to NEST will be censored at the date of the last patient visit before the study end date.
Number of adverse events as assessed by CTCAE v4.0 | 60 months
  Number of adverse events as assessed by CTCAE v4.0
Number of acute side-effects | from enrollment until 6 months after the last dose of SABR
  Acute side-effects
Number of Late side-effects | from the 6 months after the last dose of SABR until up to 3 years after inclusion in the trial
  Late side-effects
questionnaire QLQ-C30 | 60 months
  Quality of life (QoL): QoL will be evaluate with the questionnaire QLQ-C30

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria di Negrar, Negrar, Verona, Italy

IPD SHARING:
Plan to Share IPD: No